CLINICAL TRIAL: NCT01926301
Title: Cerebrovascular Autoregulation in Patients With Severe Sepsis and Septic Shock, Influence of Renal Replacement Therapy
Brief Title: Cerebrovascular Autoregulation in Sepsis, Influence of Renal Replacement Therapy
Acronym: SepsAR2
Status: Withdrawn | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Patrick Schramm, Associate Professor, Johannes Gutenberg University Mainz
Other Study IDs: 83743712
Record Dates: First submitted 2013-08-17; First posted 2013-08-20 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: sepsis; cerebrovascular autoregulation; delirium
MeSH Terms: conditions — Sepsis; Shock, Septic; Delirium | interventions — Continuous Renal Replacement Therapy; Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis: Patients with severe sepsis or septic shock with acute renal failure and requirement of continuous veno-venous hemodialysis
  Interventions: Procedure: continuous veno-venous hemodialysis
- No hemodialysis: Patients with severe sepsis or septic shock without acute renal failure and no requirement of continuous veno-venous hemodialysis

INTERVENTIONS:
Procedure: continuous veno-venous hemodialysis
  Other Names: Renal replacement therapy
  Groups: Hemodialysis

SUMMARY:
The cerebrovascular autoregulation is impaired in patients with severe sepsis and septic shock. A continuous veno-venous hemodialysis may improve impaired cerebrovascular autoregulation.

Hypothesis: continuous hemodialysis recovers impaired cerebrovascular autoregulation in patients with acute severe sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

* severe sepsis or septic shock
* adult patients
* possibility of transcranial Doppler ultrasound

Exclusion Criteria:

* traumatic brain injury
* known cerebrovascular diseases
* Infection of the brain
* chronic renal failure
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis or septic shock at the intensive care unit of an university general hospital
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular autoregulation | during the first 4 days
  Cerebrovascular autoregulation measured daily at the first 4 days of severe sepsis and septic shock

SECONDARY OUTCOMES:
Delirium | at day 4
  Incidence of Delirium at day 4 after severe sepsis or septic shock

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schramm, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- University Medical Center of the Johannes Gutenberg-Univerity, Mainz, Germany